CLINICAL TRIAL: NCT06105255
Title: A Phase I Study to Evaluate the Effects of Multiple-dose D-1553 on Pharmacokinetics of Single-dose Midazolam, Caffeine, Rosuvastatin, Furosemide and Digoxin, and to Evaluate the Effects of Multiple-dose Itraconazole and Omeprazole on Pharmacokinetics of Single-dose D-1553 in Healthy Male Subjects
Brief Title: A Study to Evaluate the Effects of D-1553 on PK of Midazolam, Caffeine, Rosuvastatin, Furosemide, Digoxin, and Itraconazole or Omeprazole on PK of D-1553
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D1553-107
Record Dates: First submitted 2023-10-17; First posted 2023-10-27 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Male

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Multipledose D-1553 on PK of single dose midazolam, caffeine, rosuvastatin, furosemide, digoxin (Experimental): To evaluate the effects of multiple-dose D-1553 tablets on pharmacokinetics (PK) of single-dose midazolam, caffeine, rosuvastatin, furosemide, and digoxin in healthy male subjects.
  Interventions: Drug: D-1553
- Evaluate the effects of multiple-dose itraconazole on PK of single-dose D-1553 (Experimental): To evaluate the effects of multiple-dose itraconazole on PK of single-dose D-1553 tablets in healthy male subjects.
  Interventions: Drug: D-1553
- Evaluate the effects of multiple-dose omeprazole on PK of single-dose D-1553 (Experimental): To evaluate the effects of multiple-dose omeprazole on PK of single-dose D-1553 tablets in healthy male subjects.
  Interventions: Drug: D-1553

INTERVENTIONS:
Drug: D-1553 — D-1553 is a novel, targeted KRASG12C inhibitor.
  Other Names: other

SUMMARY:
This is a phase I study to evaluate drug-drug interactions (DDIs) of D-1553 as a perpetrator combined with midazolam (CYP3A4 substrate), caffeine (CYP1A2 substrate), rosuvastatin (OATP1B1/OATP1B3 substrate), furosemide (OAT1/OATP1B3 substrate), and digoxin (P-gp substrate) and to evaluate DDIs of D-1553 as a victim combined with itraconazole (inhibitor of CYP3A4 and P-gp) and omeprazole (proton-pump inhibitor) in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who volunteer to participate in this clinical trial, understand the study procedures and sign the Informed Consent Form (ICF) in writing.
* Male, aged 18-45 years (both inclusive) at the time of signing the ICF.
* Non-smokers or subjects who smoked no more than 5 cigarettes or 1 pipe per day within 3 months prior to screening.

Exclusion Criteria:

* Subjects with any clinically significant acute diseases as judged by the investigators within one month prior to screening.
* Subjects who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or Treponema pallidum antibody.
* Subjects with a history of blood or needle phobia.
* Subjects with a history of hypersensitivity to the investigational drug and/or any preparation ingredients.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-24 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin: maximum concentration (Cmax). | Before and after co-administration of D-1553, approximately day1 and day10
  Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin before and after co-administration of D-1553 tablets: maximum concentration (Cmax).
Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin: area under the concentration-time curve from the time of dosing to time t (AUC0-t). | Before and after co-administration of D-1553, approximately day1 and day10
  Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin before and after co-administration of D-1553 tablets: area under the concentration-time curve from the time of dosing to time t (AUC0-t).
Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin: area under the concentration-time curve from time 0 to infinity (AUC0-∞). | Before and after co-administration of D-1553, approximately day1 and day10
  Primary PK parameters of midazolam, caffeine, rosuvastatin, furosemide, and digoxin before and after co-administration of D-1553 tablets: area under the concentration-time curve from time 0 to infinity (AUC0-∞).
Primary PK parameters of D-1553: maximum concentration (Cmax). | Before and after co-administration of itraconazole, approximately day1 and day9
  Primary PK parameters of D-1553 before and after co-administration of itraconazole: maximum concentration (Cmax).
Primary PK parameters of D-1553: area under the concentration-time curve from the time of dosing to time t (AUC0-t). | Before and after co-administration of itraconazole, approximately day1 and day9
  Primary PK parameters of D-1553 before and after co-administration of itraconazole: area under the concentration-time curve from the time of dosing to time t (AUC0-t).
Primary PK parameters of D-1553: area under the concentration-time curve from time 0 to infinity (AUC0-∞). | Before and after co-administration of itraconazole, approximately day1 and day9
  Primary PK parameters of D-1553 before and after co-administration of itraconazole: area under the concentration-time curve from time 0 to infinity (AUC0-∞).
Primary PK parameters of D-1553: maximum concentration (Cmax). | Before and after co-administration of omeprazole, approximately day1 and day8
  Primary PK parameters of D-1553 before and after co-administration of omeprazole: maximum concentration (Cmax).
Primary PK parameters of D-1553: area under the concentration-time curve from the time of dosing to time t (AUC0-t). | Before and after co-administration of omeprazole, approximately day1 and day8
  Primary PK parameters of D-1553 before and after co-administration of omeprazole: area under the concentration-time curve from the time of dosing to time t (AUC0-t).
Primary PK parameters of D-1553: area under the concentration-time curve from time 0 to infinity (AUC0-∞). | Before and after co-administration of omeprazole, approximately day1 and day8
  Primary PK parameters of D-1553 before and after co-administration of omeprazole: area under the concentration-time curve from time 0 to infinity (AUC0-∞).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui District Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No